CLINICAL TRIAL: NCT00946985
Title: A Prospective, Randomized, Active-controlled, Rater-blinded Study of the Prevention of Relapse Comparing Paliperidone Palmitate With Oral Risperidone in Adults With Recently-Diagnosed Schizophrenia Who Are at High Risk of Relapse
Brief Title: 28-30 Month Study Comparing Paliperidone Palmitate With Oral Risperidone for Treating Adults Diagnosed With Schizophrenia Within the Past 5 Years
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: The recruitment rate for the study was inadequate to achieve its enrollment goals.
Sponsor: Ortho-McNeil Janssen Scientific Affairs, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CR015646; R092670SCH3004 (Other: Ortho-McNeil Janssen Scientific Affairs, LLC)
Record Dates: First submitted 2009-07-02; First posted 2009-07-27 (Estimated); Results first posted 2012-07-16 (Estimated); Last update posted 2012-09-10 (Estimated); Status verified 2012-09

CONDITIONS: Schizophrenia
Keywords: Schizophrenia; Risperidone; Risperdal; Paliperidone Palmitate; Invega Sustenna
MeSH Terms: conditions — Schizophrenia | interventions — Paliperidone Palmitate; Risperidone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 001 (Experimental): paliperidone palmitate 50 75 100 or 150 mg eq. monthly injection for 2 years
  Interventions: Drug: paliperidone palmitate
- 002 (Active Comparator): oral risperidone 2 4 6 or 8 mg tabs once daily for two years
  Interventions: Drug: oral risperidone

INTERVENTIONS:
Drug: paliperidone palmitate — 50, 75, 100, or 150 mg eq. monthly injection for 2 years
  Arms: 001
Drug: oral risperidone — 2, 4, 6, or 8 mg tabs once daily for two years
  Arms: 002

SUMMARY:
The study will assess the use of paliperidone palmitate compared with oral risperidone in delaying time to relapse in patients recently diagnosed with schizophrenia who are at high risk of relapse.

DETAILED DESCRIPTION:
This is a Prospective, Randomized, Active-controlled, Rater-blinded Study to to assess the efficacy of paliperidone palmitate compared with oral risperidone in delaying time to relapse in patients recently diagnosed with schizophrenia who are at high risk of relapse. Recently diagnosed is defined as first diagnosis of any psychotic disorder within 5 years prior to screening. High risk of relapse is defined as having documented occurrence of 3 periods of breakthrough symptoms that required a change in patient care per the investigator's judgment (e.g., increase in dose, addition of a new drug, increase in the level of psychiatric care, notable increases in the frequency or intensity of patient contact required to maintain outpatient status, psychiatric hospitalization, etc.) within the previous 24 months, including 1 such period within the previous 6 months. Safety evaluations will include Adverse Event (AE) reporting, hematology and clinical chemistry laboratory tests, vital signs, electrocardiogram (ECG), and evaluations of suicidality and sexual functioning. Patients will receive either paliperidone palmitate 50, 75, 100, or 150 mg eq. monthly by injection for two years or oral risperidone 2, 4, 6, or 8 mg tabs once daily for two years.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be, in the opinion of the investigator, able to understand the informed consent form approved by the Institutional Review Board (IRB) or Independent Ethics Committee (IEC), as appropriate
* All patients must sign the study informed consent document indicating that they understand the purpose of and procedures required for the study and are willing to participate in the study
* Must have a current diagnosis of schizophrenia
* must have had 3 periods of breakthrough symptoms that required a change in patient care as determined by the investigator (e.g. increase in dose, addition of a new drug, hospitalization, increase in the level of psychiatric care, notable increases in the frequency or intensity of patient contact required to maintain outpatient status, etc.) within the previous 24 months, including 1 such period within the previous 6 months
* Women must be postmenopausal, surgically sterile, or otherwise be incapable of pregnancy, abstinent, or if sexually active, be practicing a highly effective method of birth control before entry, and must agree to continue to use the same method of contraception throughout the study
* Women of childbearing potential must have a negative urine pregnancy test at screening
* Patients must be cooperative and reliable, agree to receive regular injections, and be willing/able to adhere to the prohibitions and restrictions specified in this protocol.

Exclusion Criteria:

* Patients who are unable to provide their own consent or are involuntarily committed to psychiatric hospitalization
* Have attempted suicide within 12 months before screening or are at imminent risk of suicide or violent behavior
* Have a positive urine drug screen test for barbiturates, cocaine, amphetamines, or opiates at screening
* Patients who are in their first episode of psychosis
* Patients currently meeting criteria for any other Axis I diagnosis except substance abuse or an Axis II diagnosis of Mental Retardation or Borderline Personality Disorder
* Meet the Diagnostic and Statistical Manual of Mental Health Disorders fourth edition (DSM-IV) definition of substance dependence (except for nicotine and caffeine dependence) within 6-months prior to entry
* Patients with known allergies, hypersensitivity (anaphylaxis-type reaction), or intolerance to paliperidone palmitate, risperidone, Risperdal®, Risperdal® Consta®, or INVEGA® or its excipients
* Patients who received Long Acting Therapy (LAT) treatment within 2 injection cycles prior to screening
* Women who are pregnant or breast-feeding, or planning to become pregnant.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 163 (Actual)
Dates: Start 2009-06; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ortho-McNeil Janssen Scientific Affairs, LLC Clinical Trial, Study Director — Ortho-McNeil Janssen Scientific Affairs, LLC
Locations (72):
- United States (23):
  - Little Rock, Arkansas
  - Garden Grove, California
  - San Diego, California
  - Washington D.C., District of Columbia
  - Kissimmee, Florida
  - Tampa, Florida
  - Chicago, Illinois
  - Hoffman Estates, Illinois
  - Kingsport, Indiana
  - Lake Charles, Louisiana
  - Shreveport, Louisiana
  - Pittsfield, Massachusetts
  - Minneapolis, Minnesota
  - Flowood, Mississippi
  - Creve Coeur, Missouri
  - St Louis, Missouri
  - Omaha, Nebraska
  - Brooklyn, New York
  - Middleburg Heights, Ohio
  - Arlington, Texas
  - Austin, Texas
  - Irving, Texas
  - Portsmount, Virginia
- Brazil (3):
  - Curitiba
  - Salvador
  - São Paulo
- Bulgaria (3):
  - Kazanlak
  - Pleven
  - Radnevo
- Canada (5):
  - Calgary, Alberta
  - Halifax, Nova Scotia
  - Greater Sudbury, Ontario
  - Montreal, Quebec
  - Québec, Quebec
- China (8):
  - Baoding
  - Beijing
  - Changsha
  - Guangzhou
  - Kunming
  - Shanghai
  - Wuhan
  - Xi'an
- Bogotá, Colombia
- Czechia (4):
  - Kutná Hora
  - Olomouc
  - Prague
  - Strakonice
- India (9):
  - Ahmedabad
  - Aurangabad
  - Calicut
  - Hyderabad
  - Jaipur
  - Lucknow Gpo
  - Mangalore
  - Pune
  - Varanasi
- Malaysia (2):
  - Johor Bahru
  - Kuala Lumpur
- Russia (5):
  - Moscow
  - Nizny Novgorod
  - Saint Petersburg
  - Samara
  - Yaroslavl
- South Korea (4):
  - Gwangju
  - Gyeonggi-do
  - Jeonju
  - Seoul
- Ukraine (5):
  - Kharkiv
  - Kherson
  - Kiev
  - Odesa
  - Simferopol

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This trial was intended to recruit patients from multiple sites in North America, Europe, and Asia.
Pre-assignment Details: Eligible patients were to be treated with paliperdione palmitate for up to 25 weeks (stabilization phase). Patients meeting stabilization criteria were to be randomized to either paliperidone palmitate or oral risperidone and be treated for 24 months (relapse prevention phase).
Groups:
- Paliperidone Palmitate: 50, 75, 100, or 150 mg equivalent (eq.) monthly injection
Period: Stabilization Phase (25 Weeks)
Arm/Group | Paliperidone Palmitate
Started | 162
Completed | 2
Not Completed | 160
Not completed — Adverse Event | 4
Not completed — Lack of Efficacy | 3
Not completed — Lost to Follow-up | 5
Not completed — Withdrawal by Subject | 4
Not completed — Study Closed by Sponsor | 139
Not completed — Failed to Meet Stability Criteria | 2
Not completed — Prohibited Medication During Study | 1
Not completed — Patient Moved Away | 2
Period: Relapse Prevention Phase (24 Months)
Arm/Group | Paliperidone Palmitate
Started | 2 (Both randomized patients were discontinued when the sponsor terminated the trial early.)
Completed | 0
Not Completed | 2
Not completed — Study Closed by Sponsor | 2

BASELINE CHARACTERISTICS:
Arm/Group | Paliperidone Palmitate
Number analyzed (Participants) | 162
Age Continuous [Mean (Standard Deviation); unit: years] | 27 (4.55)
Age, Customized [Number; unit: participants]
  18-23 years | 46
  24-29 years | 62
  30-35 years | 54
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 54
  Male | 108
Positive and Negative Syndrome Scale (PANSS) Total Score [Mean (Standard Deviation); unit: units on a scale] — Assesses the positive symptoms, negative symptoms, and general psychopathology specifically associated with schizophrenia. The scale consists of 30 items. Each item is rated on a scale from 1 (symptom not present) to 7 (symptoms extremely severe). Scores for PANSS positive and negative each range from 7 to 49. Scores for General Psychopathology range from 16 to 112. The sum of all 30 items is defined as the PANSS total score and ranges from 30 to 210.
  units on a scale | 85.9 (13.65)
Clinical Global Impression of Severity (CGI-S) [Mean (Standard Deviation); unit: units on a scale] — The Clinical Global Impression - Severity of Illness (CGI-S) is a clinician-rated subscale (low=0, high=7, higher score indicates increasing illness). The clinician rates the severity of symptoms in relation to the clinician's total experience with schizophrenia subjects using a 7-point scale (1=normal, not at all ill, 2= borderline ill, 3= mildly ill, 4=moderately ill, 5= markedly ill, 6= severely ill, 7= among the most extremely ill subjects) in response to the question "Considering your total clinical experience with this particular population, how ill is the subject at this time?".
  units on a scale | 4.4 (0.56)
Age at First Diagnosis of Schizophrenia [Mean (Standard Deviation); unit: years] | 24.1 (4.61)
Current Schizophrenia Diagnosis [Number; unit: participants] — Per the Diagnostic and Statistical Manual for Mental Disorders fourth edition (DSM-IV) criteria.
  participants
    Paranoid (295.30) | 142
    Disorganized (295.10) | 6
    Undifferentiated (295.90) | 13
    Residual (295.60) | 1

OUTCOME MEASURES:

1. Primary Outcome: Time to Relapse During Relapse Prevention Phase
Description: Time to relapse during the relapse prevention phase was the primary efficacy variable of the study. Each case of potential relapse event were to be reviewed in a blinded fasion by an independent Relapse Monitoring Board, comprised of experts in the diagnostic, clinical and therapeutic management of schizophrenia.
Time Frame: 24 months
Population: The analysis population was to include all randomized patients who took at least one dose of study medication (ITT population). However, due to early study termination, only 2 patients were randomized and they did not have sufficient follow up. Hence the planned efficacy analysis could not be carried out.
Arm/Group | Paliperidone Palmitate
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | Paliperidone Palmitate
Serious Adverse Events (participants affected / at risk) | 6/162
Other Adverse Events (participants affected / at risk) | 50/162
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Paliperidone Palmitate (N=162)
Schizophrenia (Psychiatric disorders) | 4
Aggression (Psychiatric disorders) | 1
Depression (Psychiatric disorders) | 1
Self Injurious Behaviour (Psychiatric disorders) | 1
Hand Fracture (Injury, poisoning and procedural complications) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Paliperidone Palmitate (N=162)
Insomnia (Psychiatric disorders) | 10
Agitation (Psychiatric disorders) | 8
Anxiety (Psychiatric disorders) | 8
Restlessness (Psychiatric disorders) | 4
Headache (Nervous system disorders) | 8
Tremor (Nervous system disorders) | 8
Akathisia (Nervous system disorders) | 5
Injection Site Pain (General disorders) | 10
Weight Increased (Investigations) | 8
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 5

LIMITATIONS AND CAVEATS:
No efficacy analysis was performed due to early termination of the study (only 2 patients were randomized at the time of study termination).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No